CLINICAL TRIAL: NCT00595335
Title: Phase 2/3 Study of Rituximab for Graves' Ophthalmopathy
Brief Title: Trial of Rituximab for Graves' Ophthalmopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rebecca Bahn (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Rebecca Bahn, Professor of Medicine, Consultant in Endocrinology, Mayo Clinic, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-006130; R01DK077814-01 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2008-01-01; First posted 2008-01-16 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Thyroid-associated Ophthalmopathy
Keywords: Thyroid-associated ophthalmopathy; Rituximab; Proptosis
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos | interventions — Rituximab; Sodium Chloride; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Rituximab 1000 mg IV twice at 2-week intervals, each preceded by Methylprednisolone 100 mg IV as premedication to the rituximab infusion.
  Interventions: Drug: Rituximab; Drug: Methylprednisolone
- Placebo (Placebo Comparator): Subjects will receive 2 infusions of saline IV, 2 weeks apart, each preceded by a premedication saline IV.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Rituximab — Subjects will receive 2 infusions of rituximab (1000 mg IV), two weeks apart.
  Other Names: Rituxan; MabThera
  Arms: Rituximab
Drug: Saline — Subjects will receive 2 infusions of saline IV, 2 weeks apart, each preceded by a premedication saline IV.
  Arms: Placebo
Drug: Methylprednisolone — Subjects will receive methylprednisolone 100 mg IV as premedication to the rituximab infusion.
  Other Names: Medrol; Solu-Medrol
  Arms: Rituximab

SUMMARY:
This study is being done to investigate the effects (good and bad) of Rituximab for the treatment of an autoimmune eye disease called Graves' ophthalmopathy. This disease has proven to be difficult to treat. Rituximab is a monoclonal antibody that depletes a line of cells involved in the autoimmune response. The study hypotheses is that rituximab is effective in the treatment of patients with moderate to severe active Graves' ophthalmopathy.

DETAILED DESCRIPTION:
Laboratory evidence suggests that autoantibodies targeting the thyrotropin receptor are directly involved in the pathogenesis of Graves' ophthalmopathy (GO). This double-blind, randomized, controlled study will determine whether rituximab, an anti-B-lymphocyte antigen (CD20) monoclonal antibody that induces transient B-cell depletion, is an effective treatment for moderate to severe, active GO.

Before any treatment is given, careful eye and thyroid physical examinations will be performed and the patients will have several thyroid blood tests, a test to count the white cells in the blood, and a CT scan of the head and eyes. A close-up photograph of the face will be taken and patients will be given a short questionnaire about how their eyes are feeling and how the eye disease is affecting their quality of life.

Each study subject will receive either 2 infusions of rituximab (each 1000 mg; given 2 weeks apart) or 2 intravenous infusions of saline. Glucocorticoids (methylprednisolone 100 mg) or saline will also be administered IV as premedication to the rituximab and placebo arm respectively, in a blinded fashion but matching the randomization, to decrease the rate of infusion-associated reactions. All antihypertensive medications will be held for the 12 hours prior to and during the infusion. Patients will return 2 weeks after the first intravenous infusion in order to receive the second infusion.

Patients will be assessed at weeks 8, 16, 24 and 52 for eye disease severity, CAS, thyroid stimulating hormone (TSH), free thyroxine (fT4), free triiodothyronine (fT3), thyroid autoantibodies (TRAB), thyroid peroxidase (TPO) and C19+B cell count. CT scan of the orbits will be obtained at baseline and week 52 for orbital volume measurements and proptosis. Thyroid ultrasound will be obtained at baseline, week 24 and week 52 for thyroid volume measurements and color Doppler flow assessment.

Data analysis - Continuous variables were compared between the two treatment groups using t test or the Wilcoxon rank sum test, while categorical variables were analyzed using the chi-square /Fisher exact test. Non-parametric methods were used throughout where normality and chi-squared assumptions did not hold. General linear models were used to access treatment effect on change in CAS between baseline and 24 or 52 weeks. Patients who discontinued the trial prior to week 52 were evaluated before discontinuation and those data were carried forward to either 24 weeks (for the 5 patients who discontinued prior to or at week 24) or 52 weeks (for the single patient discontinued from the trial after 24 weeks) as the final evaluation for that patient. A p-value < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical activity score (CAS) of ≥4 and moderate to severe disease severity, as defined by thyroid eye disease severity scale based on the first letter of the defining characteristic of each class, the classification is known as: 'no signs or symptoms; only signs; soft tissue; proptosis; extraocular muscle; cornea; sight loss' (NOSPECS) score
* Euthyroid for at least 6-8 weeks
* No immediate need for decompression surgery
* With disease progression over the previous 1-2 months or without evident improvement in the prior 6 months.

Exclusion Criteria:

* Corticosteroid use in the preceding 4 weeks
* HIV, hepatitis C or hepatitis B infections
* Denied consent for HIV or hepatitis testing
* Mild or inactive Graves' ophthalmopathy
* Orbital radiotherapy within 18 months or orbital surgery within the past year
* Absolute neutrophil count < 1,500/mm^3
* Pregnant or nursing patients
* Coronary artery disease, congestive heart failure, significant arrhythmias, significant infection or immunodeficiency, other serious illnesses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Bahn, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Stan MN, Garrity JA, Carranza Leon BG, Prabin T, Bradley EA, Bahn RS. Randomized controlled trial of rituximab in patients with Graves' orbitopathy. J Clin Endocrinol Metab. 2015 Feb;100(2):432-41. doi: 10.1210/jc.2014-2572. Epub 2014 Oct 24. PMID 25343233

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Rituximab 1000 mg IV twice at 2-week intervals, each preceded by Methylprednisolone 100 mg IV as premedication to the rituximab infusion. All subjects will be treated with an acetaminophen tablet and a diphenhydramine hydrochloride tablet before the infusion.
  Rituximab: Subjects will receive 2 infusions of rituximab (1000 mg IV), two weeks apart.
  Methylprednisolone: Subjects will receive methylprednisolone 100 mg IV as premedication to the rituximab infusion.
- Placebo: Subjects will receive 2 infusions of saline IV, 2 weeks apart, each preceded by a premedication saline IV. All subjects will be treated with an acetaminophen tablet and a diphenhydramine hydrochloride tablet before the infusion.
  Saline: Subjects will receive 2 infusions of saline IV, 2 weeks apart, each preceded by a premedication saline IV.
Period: Baseline to Six Months
Arm/Group | Rituximab | Placebo
Started | 13 | 12
Completed | 11 | 10
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease Progression | 1 | 1
Not completed — Adverse Event | 1 | 0
Period: Six Months to Twelve Months
Arm/Group | Rituximab | Placebo
Started | 11 | 10
Completed | 10 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.7) | 61.8 (11.0) | 58.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Clinical Activity Score [Mean (Standard Deviation); unit: units on a scale] — The CAS, which is based on classical signs of inflammation (pain, redness, and swelling), consists of 7 equally weighted items. The total CAS (as used in this study) may range from 0 to 7. The higher the CAS, the greater degree of inflammation is present. A drop in CAS of 2 or more points suggests an improvement in the inflammatory components of the disease. A CAS ≥3 implies active disease.
  units on a scale | 4.9 (1.0) | 5.3 (1.0) | 5.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Activity Score (CAS)
Description: The clinical activity score (CAS), for Grave's ophthalmopathy has become a widely accepted tool to assess disease activity and help decide the management of the condition. The CAS, which is based on classical signs of inflammation (pain, redness, and swelling), consists of 7 equally weighted items. The total CAS (as used in this study) may range from 0 to 7. The higher the CAS, the greater degree of inflammation is present. A drop in CAS of 2 or more points suggests an improvement in the inflammatory components of the disease. A CAS ≥3 implies active disease.
Time Frame: baseline, 6 months after the first infusion
Population: Sample size was computed based on the expected drop of 2.9 and 1.5 points in the CAS score in rituximab and placebo groups. A sample size of 15 in each group will have 80% power to detect a difference in mean values of 1.4 assuming that the common standard deviation is 1.27 using a two group t-test with a 0.050 two-sided significance level.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | -1.2 (2) | -1.5 (1.8)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of the change between the two groups' CAS score at 6 months; Test type: Superiority or Other; p = 0.73, t-test, 2 sided

2. Secondary Outcome: Failure Rate
Description: The failure rate was defined as a composite variable of CAS decrease of < 2 points or need for additional therapy (excluding cosmetic surgery) for the eye disease.
Time Frame: 6 months after first infusion, 12 months after first infusion
Population: Analysis was intent to treat. The last observation was carried forward from the subjects who dropped out before (or at) 24 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
percentage of participants
  Failure rate at 6 months | 69 | 75
  Failure rate at 12 months | 46 | 50
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of the change between the two groups' failure rate at 6 months; Test type: Superiority or Other; p = 0.75, Fisher Exact
Statistical Analysis 2: Comparison: Rituximab vs Placebo; Comparison of the change between the two groups' failure rate at 12 months; Test type: Superiority or Other; p = 0.85, Fisher Exact

3. Secondary Outcome: Change in Disease Severity
Description: Disease severity was measured by the NOSPECS Score. This classification scheme of the eye changes in thyroid eye disease was introduced by the American Thyroid Association. It separates patients into seven classes of disease (class 0-6), with 0 being no signs or symptoms and 6 being sight loss. (The acronym is based on the first letter of the defining characteristic of each class, the classification is known as: 'no signs or symptoms; only signs; soft tissue; proptosis; extraocular muscle; cornea; sight loss' (NOSPECS) ).
Time Frame: baseline, 6 months after first infusion
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
participants
  Improvement by 1 class | 6 | 8
  Improvement by 2 classes | 2 | 2
  Deterioration | 2 | 0
  No change | 3 | 2

4. Secondary Outcome: Change in Proptosis
Description: Eye proptosis is a condition resulting in forward displacement of the globe from its normal position within the orbit. It is measured by computed tomography. Improvement in proptosis was defined as a decrease in proptosis by ≥2 mm.
Time Frame: baseline, 12 months after first infusion
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
mm
  Proptosis right eye | 0.82 (1.4) | 0.80 (1.3)
  Proptosis left eye | 0.1 (1.2) | 0.0 (1.8)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of the change between the two groups in proptosis in the right eye at 12 months; Test type: Superiority or Other; p = 0.97, t-test, 2 sided
Statistical Analysis 2: Comparison: Rituximab vs Placebo; Comparison of the change between the two groups in change in proptosis in left eye at 12 months; Test type: Superiority or Other; p = 0.86, t-test, 2 sided

5. Secondary Outcome: Change in Lid Fissure
Description: The palpebral fissure is the elliptic space between the medial and lateral canthi of the two open eye lids. In adults, this measures about 10mm vertically and 30mm horizontally. The fissure may be increased in vertical height in Graves' disease.
  Improvement was defined as a decrease in lid aperture width by ≥3 mm.
Time Frame: baseline, 6 months after first infusion
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
mm
  Lid fissure right eye | 0 [-1 to 1] | 0 [-1 to 1]
  Lid fissure left eye | 0 [-1.5 to 1] | 0.5 [-1 to 1.75]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of the change in lid fissure in the right eye between the two groups; Test type: Superiority or Other; p = 0.98, t-test, 2 sided
Statistical Analysis 2: Comparison: Rituximab vs Placebo; Comparison of the change in lid fissure in the left eye between the two groups; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

6. Secondary Outcome: Change in Extraocular Motility
Description: Change extraocular motility was assessed using the Gorman diplopia score. Diplopia, commonly known as double vision, is the simultaneous perception of two images of a single object that may be displaced horizontally, vertically, or diagonally (i.e., both vertically and horizontally) in relation to each other. It is usually the result of impaired function of the extraocular muscles, where both eyes are still functional but they cannot converge to target the desired object.
  The Gorman diplopia score includes four categories: 1) no diplopia (absent), 2) diplopia when the patient is tired or awakening (intermittent), 3) diplopia at extremes of gaze (inconstant), and 4) continuous diplopia in the primary or reading position (constant).
Time Frame: baseline, 6 months after first infusion, 12 months after first infusion
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale
  Change baseline-6 months | 3 [2 to 3.5] | 2.5 [0 to 4]
  Change baseline-12 months | 2 [0.75 to 3.25] | 1.5 [0.75 to 3.0]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of change between groups in extraocular motility at 6 months; Test type: Superiority or Other; p = 0.21, t-test, 2 sided
Statistical Analysis 2: Comparison: Rituximab vs Placebo; Comparison of change between groups in extraocular motility at 12 months; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

7. Secondary Outcome: Graves' Ophthalmopathy Quality of Life Score Using the Short Form-12 (SF-12) Health Survey
Description: Quality of life (QoL) was measured by the SF-12 questionnaire. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. Physical and Mental Health Composite Scores are computed (combined, scored, and weighted) using the scores of the 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Improvement was defined as a change of ≥ 6 points.
Time Frame: baseline, 6 months after first infusion, 12 months after first infusion
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale
  Baseline QoL physical | 53.2 [42.1 to 56.7] | 39.9 [33.5 to 48.8]
  Baseline QoL mental | 44.3 [32.8 to 50.7] | 46.1 [36 to 51.3]
  6 months QoL physical | 45.9 [43.6 to 50.8] | 40.3 [38.5 to 52.1]
  6 months QoL mental | 52.8 [36.1 to 56.7] | 46.1 [35.4 to 57.4]
  12 months QoL physical | 51.8 [49.8 to 55.5] | 46.7 [41.1 to 53.6]
  12 months QoL mental | 56.1 [42.8 to 57.8] | 49.4 [35.4 to 56.1]
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of the arms for QoL SF-12 physical score at 6 months; Test type: Superiority or Other; p = 0.36, t-test, 2 sided
Statistical Analysis 2: Comparison: Rituximab vs Placebo; Comparison of the arms for QoL SF-12 mental score at 6 months; Test type: Superiority or Other; p = 0.91, t-test, 2 sided
Statistical Analysis 3: Comparison: Rituximab vs Placebo; Comparison of the arms for QoL SF-12 physical score at 12 months; Test type: Superiority or Other; p = 0.29, t-test, 2 sided
Statistical Analysis 4: Comparison: Rituximab vs Placebo; Comparison of the arms for QoL SF-12 mental score at 12 months; Test type: Superiority or Other; p = 0.18, t-test, 2 sided

8. Secondary Outcome: Failure Rate at One Year
Description: as for outcome 2
Time Frame: one year
Population: Analysis was intent to treat. The last observation was carried forward from the subjects who dropped out before (or at) 52 weeks.
Measure: Number; unit: percentage of participants
Groups:
- Rituximab: Rituximab 1000 mg IV twice at 2-week intervals, each preceded by Methylprednisolone 100 mg IV as premedication to the rituximab infusion. All subjects will be treated with an acetaminophen tablet and a diphenhydramine hydrochloride tablet before the infusion.
- Placebo: Subjects will receive 2 infusions of saline IV, 2 weeks apart, each preceded by a premedication saline IV. All subjects will be treated with an acetaminophen tablet and a diphenhydramine hydrochloride tablet before the infusion.
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 13 | 12
percentage of participants | 46 | 50
Statistical Analysis 1: Comparison: Rituximab vs Placebo; Comparison of the change between the two groups' failure rate at 12 months; Test type: Superiority or Other; p = 0.85, Fisher Exact

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events for one year after the first infusion.
Arm/Group | Rituximab | Placebo
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/12
Other Adverse Events (participants affected / at risk) | 6/13 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=13) | Placebo (N=12)
Dysthroid optic neuropathy (Eye disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=13) | Placebo (N=12)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rash on face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vasculitis legs (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Significant eye tearing (Eye disorders) | 1 (1) | 0 (0)
Tongue pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis of left hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Itching of face and scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia both knees (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left eye conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No